CLINICAL TRIAL: NCT06612372
Title: Effects of 60-day-6° Head-down Bed Rest on Cartilage and Function of the Knee Joint
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M2024710
Record Dates: First submitted 2024-09-19; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Cartilage Degeneration; Weightlessness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Long term bed rest intervention group (Experimental): 60-day-6° head-down bed rest
  Interventions: Behavioral: 60-day-6° head-down bed rest

INTERVENTIONS:
Behavioral: 60-day-6° head-down bed rest — Throughout the bed rest period, subjects carried out all activities of daily living-eating, voiding, recreation, and testing

SUMMARY:
Objective: To investigate the effects of long-term simulated unloading in bed on articular cartilage quality based on functional magnetic resonance imaging (FMRI) and Knee joint function.

DETAILED DESCRIPTION:
A total of 26 subjects were recruited for a 60-day period of head-down bed rest (HDBR). The bed rest position is a 6° downward tilt of the head, and all daily activities are performed in this position. We will perform functional MRI scans of the right knee joint using T2 mapping sequences to assess tissue composition and water content before and after HDBR. Functional assessments, including the Y-Balance Test and International Knee Documentation Committee (IKDC) scores, were performed pre-HDBR and post-HDBR.We will divide each participant's knee cartilage into 18 regions and measured T2 values according to the whole organ magnetic resonance imaging score (WORMS) partitioning method.

ELIGIBILITY:
Inclusion Criteria:

* (1) male; (2) age 25-50 years old; (3) height between 160-175 cm, weight ≥50kg, and BMI between 18.5-26 kg/m²; (4) good general health status.

Exclusion Criteria:

* (1) history of alcoholism; (2) smoking ≥5 cigarettes/day in the 3 months before the test; (3) drug dependence or use of medications affecting bone metabolism within 2 weeks before screening; (4) presence of metal implants, severe vertigo, or severe snoring.

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-11-10 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
T2 mapping | three days before the HDBR started and three days after the HDBR ended
  metabolic and microstructural changes within the articular cartilage matrix components can be assessed, reflecting collagen fiber structure integrity and water content within the tissue

SECONDARY OUTCOMES:
Y-balance test | three days before the HDBR started and three days after the HDBR ended
  can comprehensively evaluate an individual's joint range of motion, lower limb strength, sense of balance, and neuromuscular control, as well as the postural control and dynamic stability of lower limbs.
International Knee Documentation Committee (IKDC) scores | three days before the HDBR started and three days after the HDBR ended
  reflects the highest level of activity that an individual is able to perform.

CONTACTS AND LOCATIONS:
Overall Officials: Jianquan Wang, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No